CLINICAL TRIAL: NCT05277558
Title: Brain Health Across the Metabolic Continuum in Youth at Risk for Type 2 Diabetes (T2D)
Brief Title: Brain Health in Youth With Normal Weight, Overweight and Obesity at Risk for Type 2 Diabetes (T2D)
Acronym: Metabrain
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202107019; 1R01DK126826-01A1 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-03-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type2 Diabetes; Type 2 Diabetes Mellitus in Obese; Dysglycemia; Microvascular Complications; Brain Structure; Obesity, Childhood; Diabetes in Adolescence; Inflammation; Insulin Resistance; Overweight, Childhood; Cognitive Decline
Keywords: Brain, Health, Youth, Type 2 Diabetes Mellitus, overweight, obesity
MeSH Terms: conditions — Pediatric Obesity; Inflammation; Insulin Resistance; Cognitive Dysfunction; Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — See page 12 of the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Weight-Normal Glucose Tolerant (NW-NGT): (1) a group that is the normal weight (BMI<85th%) and has normal glucose tolerance (NW-NGT)
  Interventions: Other: Observational
- Overweight and/or obese and has normal glucose tolerance (O-NGT): (2) a group that is overweight and/or obese (BMI >85th%) and has normal glucose tolerance (O-NGT)
  Interventions: Other: Observational
- Overweight and/or Obese and has dysglycemia (O-DG): (3) group that is overweight and/or obese (BMI >85th%) and has dysglycemia (O-DG; fasting plasma glucose ≥100 mg/dl and/or 2-hour glucose ≥140 mg/dl oral glucose tolerance test (OGTT) and laboratory-based HbA1c ≥5.8 and ≤8.0%, if treatment naïve).
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Investigators are observing brain health over time (21 months) in these groups

SUMMARY:
Investigators propose to study youth across the spectrum of body mass index (BMI) and dysglycemia. This approach will allow investigators to disentangle the relationship of key features of type 2 diabetes (T2D) risk (e.g. obesity) with intermediary physiologic changes (e.g. insulin resistance, inflammation, β-cell dysfunction and dysglycemia) that pose a risk for the brain. Investigators will determine which of these factors are most associated with differences in brain structure and function among groups, over time, and how these effects differ from normal neurodevelopment.

DETAILED DESCRIPTION:
Investigators will study three groups of pubertal youth, ages 12-17 yrs old (n=31 each): a group with normal weight and normal glucose tolerance (NW-NGT), a group with overweight/obesity and normal glucose tolerance (O-NGT), and a group with overweight/obesity and dysglycemia (O-DG). Groups will be comparable in age, sex, race/ethnicity, and socio-economic status (SES). Brain structure and function will be examined in all groups using magnetic resonance imaging (MRI) and cognitive tests at study entry (time 1/baseline), and after 21 months (time 2), focusing on a limited number of key outcome variables known to be consistently impaired in obesity or T2D. Targeted MRI measures will be regional volumes (e.g. hippocampus), neuroinflammation via restricted ratio from diffusion basis spectrum imaging (DBSI); hippocampus and white matter tracts), whole-brain cerebral blood flow via arterial spin labeling (ASL). Targeted cognitive measures will be delayed memory, processing speed, and executive function. The ultimate goal of this study is to determine how metabolic factors during neurodevelopment set the stage for the potentially profound, long-term impact of T2D on the brain and its functions. Given that the disease occurs at a time when brains are undergoing dramatic developmental processes, the aggressive nature of youth-onset T2D progression and complications in other organ systems, these results may provide guidance and justification for longer follow-up, interventional and/or mechanistic studies, and have important clinical implications.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 yrs. old at visit 1, 12-19 yrs. old at visit 2, Tanner II or above (determined through an exam by a pediatric endocrinologist or certified nurse practitioner trained in pediatric endocrinology), otherwise healthy except for obesity, <450 lbs. (due to MRI scanner limits), able and willing to lie flat within the MRI scanner and do cognitive testing, fluent in English.

Exclusion Criteria:

* Syndromic obesity, history of bariatric surgery, insulin treatment (metformin allowed if < 6 months) for T2D, contraindications for MRI (metal, claustrophobia), braces, pregnant (pregnancy test will be done on post-menarchal girls) or breastfeeding, inability to participate in cognitive testing due to sensory or language issues, intellectual disability, special education, pharmacologic treatment for Attention Deficit Hyperactivity Disorder (ADHD), prematurity (<36 weeks gestation), complications at birth, neurologic co-morbidities (e.g., seizures, stroke, head injury with >10 min loss of consciousness), significant psychiatric disorders (e.g., schizophrenia, bipolar disorder, current major depression), taking psychoactive medications (e.g., antipsychotics) that would interfere with testing or reporting illegal drug use. Self-reported smoking and alcohol use and length of time with obesity will be assessed by history (although these measures may not be fully reliable).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pubertal youth ages 12-17 yrs. will be enrolled in a longitudinal design. Investigators chose to focus on the ages where there is the highest prevalence of impaired glucose tolerance (IGT) and T2D, reducing variability in neurodevelopmental and Tanner stages in the three cohorts. Investigators will follow participants for 21 months to ensure that enough time has passed to see changes in the stated outcome measures.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
hippocampal volume | 21 months - Visit 1 and Visit 2 are 21 months apart
  To determine hippocampal volumes, investigators will use the validated, objective and semi-automatic segmentation program Automated MRI Brain Volumetry System (volBrain). Hippocampal volumes will be obtained for each subject at each visit for primary analyses. Left and right volumes will be averaged, since lateralized findings are not hypothesized.
restricted fraction | 21 months - Visit 1 and Visit 2 are 21 months apart
  Investigators will use Diffusion Basis Spectrum Imaging (DBSI) models on diffusion weighted images (DWI) to assess restricted fraction within the hippocampus and throughout white matter tracts.
Whole brain cerebral blood flow | 21 months - Visit 1 and Visit 2 are 21 months apart
  Pseudo-continuous arterial spin labeling (pCASL) will be used to measure cerebral blood flow (CBF) implemented with an arterial spin labeling (ASL) sequence 228 and volume navigators (vNavs) to minimize motion artifact. Global CBF across pairs of frames will be scaled additively to the median value. Investigators will assess the number of voxels that statistically deviate from a normative value ('distributed deviating voxels') and compared between groups.
Declarative Memory | 21 months - Visit 1 and Visit 2 are 21 months apart
  Investigators will use the total score from the Paired Associates Memory Test, an experimental cognitive task measuring delayed declarative memory
Processing speed | 21 months - Visit 1 and Visit 2 are 21 months apart
  Investigators will use the raw scores from the NIH Toolbox Pattern Comparison Processing Speed task.
Executive Function | 21 months - Visit 1 and Visit 2 are 21 months apart
  Investigators will use an average of the (z scores) from the NIH Toolbox Flanker Inhibitory Control & Attention, Dimensional Change Card Sort and List Sorting tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara A Hershey, PhD, Principal Investigator — Washington University School of Medicine; Silva Arslanian, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Investigators affirm that data and research resources will be shared. Any shared data will have low re-identification potential. The Research Design & Biostatistics Group of the investigative team's Washington University's Clinical Translational Science Award (CTSA) provides access to the REDCap database to facilitate secure data sharing with approved investigators within the University as well as with approved collaborators. De-identified MRI scans will be shared with approved investigators through the Central Neuroimaging Data Archive (CNDA), an online, secure image archive system.
Supporting Information: Study Protocol
Time Frame: within 12 months of end of data collection, data entry, quality control and image processing
Access Criteria: PI will need to request data for legitimate scientific purpose.